CLINICAL TRIAL: NCT04588597
Title: Obstetric and Neonatal Outcomes of Twin Pregnancy (Twin Conception-To-Birth): A Multicenter International Study
Brief Title: Obstetric and Neonatal Outcomes of Twin Pregnancy
Acronym: Twin-CTB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Middle-East OBGYN Graduate Education Foundation (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, M.B.B.Ch, M.S.c in Gynecology and Obstetrics, Assiut University
Other Study IDs: Twin-CTB
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Twin Pregnancy
Keywords: Twin pregnancy; maternal outcomes; neonatal outcomes; machine learning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter study aims at assessing the natural history of twin pregnancy and developing a machine learning-based algorithm to predict clinical outcomes of twin pregnancy during pregnancy and delivery and to determine management strategies that are associated with best maternal and neonatal outcomes. This study will include at least 12 centers from different countries that present at least Europe, South America, Asia, and Africa. Data will be retrospectively collected from January 1st, 2010 to December 31st, 2019.

DETAILED DESCRIPTION:
Twin pregnancies carry higher risks of maternal, fetal and neonatal adverse outcomes compared to singleton pregnancy.They are associated with increased perinatal morbidity and mortality, anemia, pregnancy- induced hypertension, increased incidence of cesarean section (CS), postpartum hemorrhage, prematurity and low birth weight and Increased rate of perinatal death.

This multicenter study aims at assessing the natural history of twin pregnancy, and developing a machine learning-based algorithm to predict clinical outcomes of twin pregnancy during pregnancy and delivery and to determine management strategies that are associated with best maternal and neonatal outcomes.

Medical records of eligible women will be reviewed, and data abstraction will be performed using a standardized excel sheet designed for this study. Target data include baseline demographics and clinical data (e.g. age, parity, ethnicity, smoking, IVF pregnancy, history of gynecologic surgeries, type of twin pregnancy, current medical disorders, current obstetric complications, fetal anomalies, administration of antenatal steroids, Placental site, and twin-specific complications). Information from serial ultrasound reports including fetal growth and Doppler studies will be collected and data on fetal intervention will be abstracted. Peripartum data include node of delivery, Method of induction, CS indication, and type of cesarean incision. Clinical outcomes include postpartum hemorrhage, and perinatal death, admission to neonatal intensive care unit (NICU), neonatal need for respiratory support, neonatal intracranial hemorrhage, neonatal respiratory distress syndrome and neonatal hypoxic ischemic encephalopathy. Data will not include any identifiable information.

Prediction model will be created using baseline demographic and obstetric features of pregnancy and individual maternal and perinatal complications will be set as outcomes (dependent variables). A composite outcome of major maternal and neonatal outcomes will be created separately.

ELIGIBILITY:
Inclusion Criteria:

1. Women with twin pregnancy who received their antenatal care and were delivered in the participating institute
2. Compliance to antenatal care visits

Exclusion Criteria:

1. Major fetal anomalies of one or both twins
2. Elective miscarriage
3. Authorization to use medical records was not provided by the patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include eligible women from at least 12 centers(anticipated) from different countries that present at least Europe, South America, Asia, and Africa.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum hemorrhage | From delivery of the baby to 24 hours postoperative (Total of 24 hours)
  Significant uterine bleeding > 1000 ml
perinatal death | From onset of labor to 1 week postnatal
  Death of the baby during delivery or early neonatal period
Admission to neonatal intensive care unit (NICU) | From delivery of the baby to 24 hours postoperative (Total of 24 hours)
  Admission of the baby to NICU for observation or intervention
Intrauterine fetal death | Death of the fetus any time from 24 weeks to onset of labor

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Shazly, M.Sc, Principal Investigator — Assiut University

REFERENCES:
- [Background] Qin JB, Wang H, Sheng X, Xie Q, Gao S. Assisted reproductive technology and risk of adverse obstetric outcomes in dichorionic twin pregnancies: a systematic review and meta-analysis. Fertil Steril. 2016 May;105(5):1180-1192. doi: 10.1016/j.fertnstert.2015.12.131. Epub 2016 Jan 19. PMID 26801066
- [Background] Huang J, Maguire MG, Ciner E, Kulp MT, Cyert LA, Quinn GE, Orel-Bixler D, Moore B, Ying GS; Vision in Preschoolers (VIP) Study Group. Risk factors for astigmatism in the Vision in Preschoolers Study. Optom Vis Sci. 2014 May;91(5):514-21. doi: 10.1097/OPX.0000000000000242. PMID 24727825
- [Background] Adinma JI, Agbai AO. Multiple births in Nigerian Igbo women: incidence and outcomes. J Obstet Gynaecol. 1997 Jan;17(1):42-4. doi: 10.1080/01443619750114077. PMID 15511763
- [Background] Mutihir JT, Pam VC. Obstetric outcome of twin pregnancies in Jos, Nigeria. Niger J Clin Pract. 2007 Mar;10(1):15-8. PMID 17668709
- [Background] Rzyska E, Ajay B, Chandraharan E. Safety of vaginal delivery among dichorionic diamniotic twins over 10 years in a UK teaching hospital. Int J Gynaecol Obstet. 2017 Jan;136(1):98-101. doi: 10.1002/ijgo.12017. Epub 2016 Nov 3. PMID 28099698
- [Background] Kong CW, To WWK. The predicting factors and outcomes of caesarean section of the second twin. J Obstet Gynaecol. 2017 Aug;37(6):709-713. doi: 10.1080/01443615.2017.1286466. Epub 2017 Mar 21. PMID 28325122
- [Background] Kato K, Fujiki K. Multiple births and congenital anomalies in Tokyo Metropolitan Hospitals, 1979-1990. Acta Genet Med Gemellol (Roma). 1992;41(4):253-9. doi: 10.1017/s0001566000002117. PMID 1342133
- [Background] Rodis JF, McIlveen PF, Egan JF, Borgida AF, Turner GW, Campbell WA. Monoamniotic twins: improved perinatal survival with accurate prenatal diagnosis and antenatal fetal surveillance. Am J Obstet Gynecol. 1997 Nov;177(5):1046-9. doi: 10.1016/s0002-9378(97)70012-7. PMID 9396891
- [Background] Carroll SG, Soothill PW, Abdel-Fattah SA, Porter H, Montague I, Kyle PM. Prediction of chorionicity in twin pregnancies at 10-14 weeks of gestation. BJOG. 2002 Feb;109(2):182-6. doi: 10.1111/j.1471-0528.2002.01172.x. PMID 11905430
- [Background] Lee YM, Cleary-Goldman J, Thaker HM, Simpson LL. Antenatal sonographic prediction of twin chorionicity. Am J Obstet Gynecol. 2006 Sep;195(3):863-7. doi: 10.1016/j.ajog.2006.06.039. PMID 16949427
- [Background] Cao K, Verspoor K, Sahebjada S, Baird PN. Evaluating the Performance of Various Machine Learning Algorithms to Detect Subclinical Keratoconus. Transl Vis Sci Technol. 2020 Apr 24;9(2):24. doi: 10.1167/tvst.9.2.24. eCollection 2020 Apr. PMID 32818085